CLINICAL TRIAL: NCT06865729
Title: Effect of Music Therapy Applied to Hospitalized Chronically Ill Individuals on Hospital Anxiety, Depression and Comfort Levels: A Randomized Controlled Trial
Brief Title: Effect of Music Therapy on Hospital Anxiety/Depression and Comfort Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Kübras, Master Student, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AUSBF-SARI-001
Record Dates: First submitted 2024-11-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group (Experimental): Music Therapy
  Interventions: Behavioral: Music therapy
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Music therapy — Music therapy will be performed by the researchers for 4 days (average length of stay for inpatients is 4 days), starting from the first day the patients start their inpatient treatment. Music therapy will be performed in the evening hours (between 20:00 and 21:00) and in the patients' own rooms, so as not to disrupt the patients' routine follow-up and treatment. Music therapy will be performed passively using an MP3 music player and headphones provided by the researchers. Therapy time will be limited to 30 minutes. Music therapy will be performed in one session per day for 4 days, and the patients will listen to the same music in each session.
  Arms: Participant Group

SUMMARY:
Aim: It has been determined that there are limited studies in our country where music is used as a nursing intervention and the effects of music therapy on the psychological symptoms and comfort levels of individuals with chronic diseases are evaluated. This study will be conducted to determine the effects of music therapy applied to hospitalized individuals with chronic diseases on hospital anxiety, depression and comfort levels.

The research will be conducted at the Urology Department of Merzifon Kara Mustafa Paşa State Hospital between September 2024 and May 2025. The research is a randomized controlled experimental type. The sample of the research will consist of 60 participants, 30 in the music therapy group and 30 in the control group, who are 18 years of age and older and diagnosed with chronic diseases.

Data in the research: The research data will be collected using the Personal Information Form, Hospital Anxiety and Depression Scale and General Comfort Scale Short Form.

In this study, music therapy will be performed by the researchers for 4 days (the average length of stay of inpatients is 4 days), starting from the first day the participants start their inpatient treatment in the hospital. The data collection forms will be applied twice in total, at the first interview (pre-test) and on the morning of the 5th day (post-test).

DETAILED DESCRIPTION:
It has been determined that anxiety and depression in individuals with chronic diseases are strongly and independently associated with mental health and physical symptom burden, and depression also has an important relationship with quality of life areas. Anxiety and depression negatively affect the continuation of treatment, its effectiveness and the quality of life of individuals in chronic diseases. All these negative situations experienced by patients also cause a decrease in comfort. Elimination or reduction of situations that disturb patients is only possible by increasing comfort. It is known that patients with a high level of comfort recover more quickly and can cope with the disease process more easily.

Various pharmacological treatments are applied to alleviate the anxiety and depression levels in individuals with chronic diseases, and these treatments have important side effects that affect the body and mind. For this reason, the use of non-pharmacological treatments such as cognitive behavioral therapy, physical activity, group therapies, relaxation and dreaming methods, aromatherapy, laughter therapy and hypnosis has become privileged in overcoming depression and anxiety in individuals with chronic diseases. Music therapy is another non-pharmacological treatment frequently used to relieve depression and anxiety.

Data analysis: The data obtained from the research will be analyzed in the Statistical Package for Social Science (SPSS) 21 statistical program. Variables covering the introductory characteristics of individuals with chronic diseases will be expressed as numbers and percentages. The Shapiro-Wilk test will determine whether the data show a normal distribution and parametric and/or non-parametric tests will be used according to the results obtained. Statistical significance will be accepted as p<.05.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Being hospitalized due to a chronic disease
* Speaking and understanding Turkish
* Not using any medication that would affect anxiety and depression
* Giving consent to participate in the study

Exclusion Criteria:

* Having been diagnosed with any psychiatric/neurological disease
* Having problems with sensory perception and communication skills

Min Age: 18 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | A pre-test will be applied after the patients are admitted to the clinic. The post-test will be applied on the 5th day of the patients' hospitalization.
  The scale was developed by Zigmond and Snaith (1983).The adaptation of the scale to Turkish and its validity and reliability analyses were conducted by Aydemir et al. in 1997.The scale consists of 14 items. Odd-numbered items investigate anxiety and even-numbered items investigate depression.The scale is a four-point Likert-type assessment tool and the scores of the items range from 0 to 3.However, each item is scored differently; items 1, 3, 5, 6, 8, 10, 11 and 13 show decreasing severity and are scored as 3, 2, 1, 0. On the other hand, items 2, 4, 7, 9, 12 and 14 are scored as 0, 1, 2, 3.The total scores of the subscales are obtained by summing the scores of these items.For the anxiety subscale, items 1, 3, 5, 7, 9, 11 and 13 are added; for the depression subscale, items 2, 4, 6, 8, 10, 12 and 14 are added.The cut-off point for the anxiety subscale of the Turkish form of the Hospital Anxiety and Depression Scale was found to be 10, and the cut-off point for the depression subscale.
Shortened General Comfort Questionnaire (SGCQ) | A pre-test will be applied after the patients are admitted to the clinic. The post-test will be applied on the 5th day of the patients' hospitalization.
  The scale was developed by Kolcaba in 2006. The Turkish validity and reliability study of the scale was conducted by Çıtlık Sarıtaş et al. (2018). The scale consists of 28 items and the items of the scale are scored between 28-168. The lowest possible value, 1, indicates low comfort, and the highest value, 6, indicates high comfort. The General Comfort Scale Short Form includes the sub-dimensions of Relief (9 items), Relaxation (9 items), and Superiority (10 items). The total score obtained is divided by the number of scale items to find the mean value. The Cronbach alpha reliability coefficient of the Turkish form of the scale was found to be 0.82. The Cronbach alpha reliability coefficients of the scale sub-dimensions (relief, relaxation, and superiority) were found to be 0.81, 0.81, and 0.76, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Sarı, MSc, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Merkez, Amasya, Turkey (Türkiye)